CLINICAL TRIAL: NCT00208455
Title: An Uncontrolled, Multi-Centre, Prospective, Post Marketing Surveillance Study to Monitor the Long Term Survivorship of the DePuy PROXIMA™ Hip in Subjects Requiring a Total Hip Replacement
Brief Title: A Multi-centre Study to Assess the Long-term Performance of the DePuy PROXIMA™ Hip in Primary Total Hip Replacement
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: DePuy discontinued this product in 2013, the clinical program was reviewed and this Study was closed.
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT03/09
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Post-traumatic Arthritis; Avascular Necrosis; Traumatic Femoral Fractures; Congenital Hip Dysplasia
Keywords: Arthroplasty; Replacement; Hip; Conservative; Anatomic; Cementless
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Osteonecrosis; Hip Dislocation, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DePuy Proxima™ Hip (Other): A short, anatomic, cementless femoral component for use in total hip arthroplasty
  Interventions: Device: DePuy Proxima™ Hip

INTERVENTIONS:
Device: DePuy Proxima™ Hip — A short, anatomic, cementless femoral component for use in total hip arthroplasty

SUMMARY:
The purpose of this study is to monitor the performance of the DePuy PROXIMA™ hip in the treatment of patients with hip joint disease requiring a total hip replacement. Patients who enter the study will be evaluated at regular intervals following hip surgery using patient, clinical and x-ray assessments. A subset of patients will undergo scans to allow the bone mineral density of the bone surrounding the implant to be monitored

ELIGIBILITY:
Inclusion Criteria:

i) Male or female subjects between 18 and 70 years of age.

ii) Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.

iii) Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and agree to return to the hospital for all the required post-operative follow-ups.

iv) Subjects who are scheduled to undergo a primary total hip replacement whom the surgeon considers to be suitable for the DePuy PROXIMA™ hip femoral prosthesis.

Exclusion Criteria:

i) Subjects who, in the opinion of the Investigator, have an existing condition/co-morbidity or infection that would compromise their long term participation and follow-up in this study.

ii) Women who are pregnant.

iii) Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.

iv) Subjects who have participated in a clinical study with an investigational product in the last 6 month(s).

v) Subjects who are currently involved in any injury litigation claims.

vi) Subjects for whom the surgical procedure is a revision of a previous THR or hemi-arthroplasty, or who have previously undergone arthrodesis or osteotomy of the hip.

vii) Subjects undergoing a simultaneous bilateral hip operation.

viii) Subjects undergoing the second stage of a staged bilateral for whom the contralateral hip is part of this clinical investigation.

ix) Subjects undergoing the second stage of a staged bilateral for whom the contralateral hip was implanted less than six months previously or is not performing satisfactorily

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2005-02; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Kaplan-Meier survivorship calculated at the five-year time-point | 5 yrs

SECONDARY OUTCOMES:
Annual Kaplan-Meier survivorship calculations | Annually
Harris Hip Score | 6mths, 1yr, 2yrs, 5yrs, 7 yrs, 10yrs and 15 yrs post-surgery
Radiographic analysis | 6mths, 1yr, 2yrs, 5yrs, 7yrs, 10yrs and 15yrs post-surgery
Oxford Hip score | 6mths, and annually post-surgery

CONTACTS AND LOCATIONS:
Locations (4):
- Asklepios Klinikum, Bad Abbach, Germany
- Ospedale San Pietro, Rome, Italy
- Arnau de Vilanova, Valencia, Spain
- North Bristol NHS Trust, Bristol, United Kingdom